CLINICAL TRIAL: NCT04773639
Title: Randomized Clinical Trial of a Multi-Modal Palliative Care Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Rocky Mountain Cancer Centers (Other); University of Colorado, Denver (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Joanna Arch, Associate Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 19-0787; R01NR018479 (NIH)
Record Dates: First submitted 2021-02-10; First posted 2021-02-26 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Depression, Anxiety; Metastatic Cancer
MeSH Terms: conditions — Depression; Anxiety Disorders; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: In a randomized controlled trial, this project evaluates the M-ACT intervention for community patients with metastatic cancer relative to the usual care control condition, reflecting Stage IIb/III of the NIH stage model for evaluating behavioral interventions. We will randomize 240 patients to M-ACT or usual care for five weeks (n per condition = 120) and assess them at Baseline (Pre), Mid-Intervention (Mid), Post-Intervention (Post), and 2-month Follow-Up (FU).
Who Masked: Investigator, Outcomes Assessor
Masking Description: The PI will be blinded to condition assignment. Outcomes will be assessed in REDCap.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-Modal Acceptance and Commitment Therapy (M-ACT) (Experimental): M-ACT consists of five 2-hour group sessions (plus booster) that alternate with self-paced online modules and check-ins that participants complete on their own, between the group sessions. The intervention addresses distress associated with coping with metastatic cancer and supports engagement in advance care planning. The intervention is based on Acceptance and Commitment Therapy, an intervention model that aims to help people cope with life challenges and difficult thoughts/feelings in a manner that helps them to live fuller and more meaningful lives.
  Interventions: Behavioral: Multi-Modal Palliative Care Intervention
- Control: Usual Care (Other): Patients in the control arm will have access to usual care (UC) at the collaborating clinics, consisting of access to a clinical social worker and nurse practitioners for advance care planning and supportive visits at patient request. After completion of study procedures, including FU, the UC participants will be offered M-ACT free of cost.
  Interventions: Behavioral: Usual Care Control Condition

INTERVENTIONS:
Behavioral: Multi-Modal Palliative Care Intervention — An innovative muli-modal palliative care intervention that addresses the lack of advance care planning and unmet psychosocial needs commonly experienced by patients with metastatic cancer.
  Arms: Multi-Modal Acceptance and Commitment Therapy (M-ACT)
Behavioral: Usual Care Control Condition — The control condition includes usual care (UC) at the collaborating clinics, consisting of access to a clinical social worker and nurse practitioners for advance care planning and supportive visits at patient request.
  Arms: Control: Usual Care

SUMMARY:
Adults diagnosed with metastatic cancer commonly experience depression and anxiety symptoms, which can interfere with advance care planning. This randomized clinical trial evaluates a novel, piloted, primary palliative care intervention that addresses advance care planning and psychosocial needs of patients with metastatic cancer. The intervention focuses on patients with elevated anxiety and depression (anx/dep) symptoms-those with highest psychosocial needs who may be at greatest risk for advance care planning non-completion. The intervention is founded on an evidence-based intervention approach known as Acceptance and Commitment Therapy (ACT) that reduces distress and promotes behavior change through theory-driven mechanisms. In the proposed randomized trial, M-ACT will be compared to a usual care control condition. The study will also assess the association between advance care planning and anx/dep symptoms, thereby informing the critical practice question of whether anx/dep symptoms should be addressed concurrently with advance care planning. The study will enroll patients with Stage IV solid tumor cancer (N=240) within Rocky Mountain Cancer Centers, randomized 1:1 to M-ACT or usual care. The study aims to: 1) Evaluate the hypothesis that M-ACT will increase advance care planning completion (primary outcome) and sense of life meaning, and reduce anx/dep symptoms and fear of dying relative to usual care control. 2) Assess the association between anx/dep symptoms and advance care planning at baseline and over time, testing the hypothesis that decreases in anx/dep symptoms at post- intervention will be associated with increases in advance care planning at follow-up. 3) Assess M-ACT's hypothesized mechanisms to specify how the intervention works (exploratory aim). Given their advance care planning and psychosocial needs, and poor access to palliative care, rigorously investigating M-ACT has the potential to benefit community patients with metastatic cancer and to advance palliative care science by addressing gaps in novel approaches, foundational knowledge, and the scalable delivery of palliative care.

Note: Due to the coronavirus pandemic, the in-person group component of M-ACT has currently been shifted to an online group format.

DETAILED DESCRIPTION:
This study will evaluate an innovative, multi-modal palliative care intervention that addresses the lack of advance care planning (ACP) and unmet psychosocial needs commonly experienced by patients with metastatic cancer. Up to half of adults with metastatic cancer report elevated anxiety or depression symptoms, which can cause withdrawal from daily activities and future planning and have been linked to non-adherent health behaviors in other disease populations. However, little is known about the extent to which anxiety or depression influence ACP completion in palliative care. In addition, metastatic cancer triggers patients' fear of dying and threatens their sense of meaning. The current approach aims to optimize two core palliative care outcomes - ACP and psychosocial well being - in outpatient oncology settings and to build the evidence base for primary palliative care interventions. This new multimodal intervention, which is based on extensive pilot data, uses a primary palliative care approach and focuses on patients with elevated anxiety or depression (anx/dep) symptoms.

The intervention is based on Acceptance and Commitment Therapy (ACT), an evidence-based approach to reduce distress and promote behavior change through theorized mechanisms that include cultivating acceptance of internal experience and aligning behavior with personal values. A pilot study for adults with metastatic cancer and elevated anx/dep symptoms conducted by the current research team, leveraged ACT to design and refine the multi-modal ACT intervention (M-ACT) in response to patient and provider feedback. M-ACT helps metastatic cancer patients to live meaningfully and face the future no matter what their health status, supports their engagement in ACP and addresses their psychosocial needs.

To facilitate future scalability, M-ACT uses a novel multi-modal delivery structure comprising both in-person group sessions led by existing on-site clinical social workers and self-paced, personalized online sessions completed at home, which efficiently increase intervention dose without increasing patient travel or provider demands. The current randomized controlled trial will rigorously evaluate the ability of M-ACT to increase ACP (primary outcome) and improve psychosocial outcomes (secondary). This study also will evaluate the relationship between anx/dep symptoms and ACP to inform the critical clinical question of whether anx/dep symptoms should be addressed concurrently with ACP. Finally, the study will explore mechanisms that may explain how M-ACT influences ACP and the targeted secondary outcomes.

The study will enroll patients with stage IV solid tumor cancer (N = 240), randomized in a 1:1 ratio to M-ACT or usual care for a 4-week intervention period. Outcomes will be assessed at baseline, mid-intervention (to assess mechanisms), 1-week post-intervention, and 2-month follow-up.

Note: Due to the coronavirus pandemic, the in-person group component of M-ACT has currently been shifted to an online group format.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. English-speaking (able to speak, read, and write well in English)
3. Diagnosed with Stage IV metastatic cancer of any solid tumor type
4. Capable at time of consent of understanding and voluntarily consenting themselves to the study, attending group sessions, and completing the online sessions at home, confirmed by an Eastern Cooperative Group Performance Status Scale of 0 to 2
5. Endorse moderate to severe anxiety or depression symptoms on the Patient Health Questionnaire-4

Exclusion Criteria:

1. Current high suicide risk
2. Psychiatric hospitalization or suicide attempt in the past 5 years
3. History of chronic, untreated trauma unrelated to their cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Change in advance care planning | Assessed four times with parallel timing in the control group: prior to the intervention (Pre), week 3 of the intervention (Mid), within one week after the end of the weekly intervention (Post), at 2-month follow-up (FU)
  The primary outcome is defined as change in the number of steps taken toward ACP completion from baseline through 2-month follow-up. ACP steps will be assessed with a checklist adapted from the M-ACT pilot study by consulting the Hospice & Palliative Nurses Association online ACP resources and the study team, and refined by soliciting pilot participants' feedback on item clarity. The checklist describes each ACP step and asks patients to indicate steps taken to date.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | Assessed four times with parallel timing in the control group: prior to the intervention (Pre), week 3 of the intervention (Mid), within one week after the end of the weekly intervention (Post), at 2-month follow-up (FU)
  Patient-reported depression symptom questionnaire. Higher scores = more depression symptoms
Generalized Anxiety Disorder-7 | Assessed four times with parallel timing in the control group: prior to the intervention (Pre), week 3 of the intervention (Mid), within one week after the end of the weekly intervention (Post), at 2-month follow-up (FU)
  Patient-reported anxiety symptom questionnaire. Higher scores = more anxiety symptoms
The Death Attitude Profile - Revised, Fear of Death and Death Avoidance Scales | Assessed four times with parallel timing in the control group: prior to the intervention (Pre), week 3 of the intervention (Mid), within one week after the end of the weekly intervention (Post), at 2-month follow-up (FU)
  Patient-reported fear of death and dying questionnaire. Higher scores = greater fear of death and dying
Functional Assessment of Chronic Illness Therapy (FACIT), Meaning/Peace Subscale | Assessed four times with parallel timing in the control group: prior to the intervention (Pre), week 3 of the intervention (Mid), within one week after the end of the weekly intervention (Post), at 2-month follow-up (FU)
  Patient-reported sense of life meaning and peace. Higher scores = greater sense of meaning/peace

OTHER OUTCOMES:
Intervention Acceptability: Session Feedback Questionnaire | At the end of each session during the 5-week intervention period, plus after the booster session 1 month later
  Participant value of the session will be assessed through the Session Feedback. Higher scores = higher value and acceptability of the session
Intervention Acceptability: Group session attendance and online session completion | From the start to end of the 5-week intervention plus the booster session held 1 month later
  Intervention engagement will be assessed via attendance in group sessions and completion of the online modules and check-ins
Intervention Acceptability: Client Satisfaction Questionnaire-8 | Assessed two times: within one week after the end of the weekly intervention (Post), at 2-month follow-up (FU)
  Participant satisfaction will be measured using the Client Satisfaction Questionnaire-8 (adapted to the current intervention) with higher scores indicating more satisfaction
Process measure: Multidimensional Experiential Avoidance Scale: Denial and Distress Aversion scales | Assessed four times with parallel timing in the control group: prior to the intervention (Pre), week 3 of the intervention (Mid), within one week after the end of the weekly intervention (Post), at 2-month follow-up (FU)
  Patient-reported experiential avoidance with higher scores indicating greater avoidance.
Process Measure: Experiences Questionnaire-Decentering Scale | Assessed four times with parallel timing in the control group: prior to the intervention (Pre), week 3 of the intervention (Mid), within one week after the end of the weekly intervention (Post), at 2-month follow-up (FU)
  Patient-reported defusion/decentering with higher scores indicating greater defusion/decentering.
Process Measure: Valuing Questionnaire | Assessed four times with parallel timing in the control group: prior to the intervention (Pre), week 3 of the intervention (Mid), within one week after the end of the weekly intervention (Post), at 2-month follow-up (FU)
  Patient-reported values-aligned behavior with higher scores indicating more aligned behavior

CONTACTS AND LOCATIONS:
Overall Officials: Joanna J Arch, PHD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Rocky Mountain Cancer Centers, Boulder, Colorado, United States

REFERENCES:
- [Background] Arch JJ, Fishbein JN, Ferris MC, Mitchell JL, Levin ME, Slivjak ET, Andorsky DJ, Kutner JS. Acceptability, Feasibility, and Efficacy Potential of a Multimodal Acceptance and Commitment Therapy Intervention to Address Psychosocial and Advance Care Planning Needs among Anxious and Depressed Adults with Metastatic Cancer. J Palliat Med. 2020 Oct;23(10):1380-1385. doi: 10.1089/jpm.2019.0398. Epub 2020 Jan 6. PMID 31905307
- [Derived] Arch JJ, Mitchell JL, Schmiege SJ, Levin ME, Genung SR, Nealis MS, Fink RM, Bright EE, Andorsky DJ, Kutner JS. A randomized controlled trial of a multi-modal palliative care intervention to promote advance care planning and psychological well-being among adults with advanced cancer: study protocol. BMC Palliat Care. 2022 Nov 17;21(1):198. doi: 10.1186/s12904-022-01087-z. PMID 36384735